CLINICAL TRIAL: NCT07109479
Title: A Prospective, Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of the Single-Use Coronary Forward Intravascular Lithotripsy Catheter Combined With the Intravascular Lithotripsy Therapy Device for Pre-treatment of De Novo Calcified Stenotic Coronary Lesion
Brief Title: Safety and Effectiveness of the Single-Use Coronary Forward Intravascular Lithotripsy Catheter Combined With the Intravascular Lithotripsy Therapy Device
Acronym: FORWARD IVL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spectrumedics Medical Technology(Shanghai)Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC-SWFC-01
Record Dates: First submitted 2025-07-22; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Coronary Arterial Disease
MeSH Terms: interventions — Atherectomy, Coronary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular Lithotripsy (Experimental)
  Interventions: Device: Intravascular Lithotripsy
- Coronary Rotational Atherectomy (Active Comparator)
  Interventions: Device: Rotational Atherectomy

INTERVENTIONS:
Device: Intravascular Lithotripsy — study group will receive the investigational devices (Single-Use Coronary Forward Intravascular Lithotripsy Catheter combined with the Intravascular Lithotripsy Therapy Device) for calcified lesion pre-treatment.
  Arms: Intravascular Lithotripsy
Device: Rotational Atherectomy — control group will receive the control device (Coronary Rotational Atherectomy System)
  Arms: Coronary Rotational Atherectomy

SUMMARY:
The FORWARD IVL trial is a Prospective, Multicenter Study conducted to assess the safety and effectiveness of the Single-Use Coronary Forward Intravascular Lithotripsy Catheter combined with the Intravascular Lithotripsy Therapy Device for the pre-treatment of calcified, stenotic de novo coronary artery lesions .

DETAILED DESCRIPTION:
The approved IVL devices are based on balloon design, and the biggest limitation is the crossability, especially in the severe stenosis lesions.

Coronary Forward IVL Catheter allow the catheter to modify calcium in tight, difficult to cross lesions to increase the compliance of the vessel and allow further crossing of the device or additional treatment.

This trial consists of two parts:

Part 1 (RCT part): this part is a prospective, multicenter, randomized controlled, study in subjects with moderate-to-severe calcification.180 eligible subjects are planned to enroll .

Part 2 (Single-arm part):This part is a single-arm study in subjects with calcified lesions that are Chronic Total Occlusions (CTOs)(with minimum 30 subjects).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* 1) Age ≥18 years, male or female.

  2)Primary coronary artery disease (with evidence of asymptomatic myocardial ischemia, stable/unstable angina, or old MI) scheduled for non-emergent PCI.

  3)Pre-procedure Left Ventricular Ejection Fraction (LVEF) ≥30%.

  4)Voluntarily participate in this study and sign Informed Consent Form (ICF), willing to comply with study procedures and follow-up.

Angiographic Inclusion Criteria:

1. Target lesion is de novo calcified stenotic coronary lesion with no prior intervention.
2. Target lesion reference vessel diameter is 2.5-4.0 mm.
3. Target lesion meets ONE of the following:

   RCT part: Moderate-to-severe calcification AND stenosis ≥90% and <100% (length ≤60 mm). (Moderate Calcification: Clearly visible high-density shadows during cardiac motion; Severe Calcification: Clearly visible high-density shadows visible without cardiac motion).

   Single-arm part: Calcified lesion AND Chronic Total Occlusion (CTO) (length ≤20 mm).
4. Guidewire positioned in the true lumen distal to the target lesion and not in the subintimal space prior to device use.

Exclusion Criteria:

General Exclusion Criteria

* 1) Planning use of scoring/cutting balloons, Excimer Laser Coronary Atherectomy (ELCA), or Coronary Intravascular Lithotripsy balloons for calcified lesion modification prior to study device use.

  2) NYHA Class III or IV.

  3) Currently on dialysis or serum creatinine level >2.5 mg/dL (or 221 µmol/L).

  4) Severe coagulation disorder (platelet count <100×10⁹/L).

  5) Hyperviscosity diseases (e.g., polycythemia vera, platelet count >750×10⁹/L).

  6) Cardiac shock with clinical signs or symptoms.

  7) Active systemic infection.

  8) Moderate-to-severe anemia (hemoglobin <90 g/L).

  9) Acute Myocardial Infarction within 1 month prior to procedure.

  10) Stroke or Transient Ischemic Attack (TIA) within 3 months prior to procedure.

  11) Active gastrointestinal ulcer or bleeding within 3 months prior to procedure.

  12) Expected life expectancy <12 months as assessed by the investigator.

  13) Known intolerance to antiplatelet or anticoagulant therapy.

  14) Known allergy to study device components or contrast media.

  15) Known pregnancy or lactation (female subjects).

  16) Participating or planning to participate in another drug or device clinical trial.

  17) Other conditions deemed unsuitable for participation by the investigator

Angiographic Exclusion Criteria:

1. Unprotected left main coronary artery disease (stenosis >50%).
2. Serious angiographic complication in the target vessel prior to study device use.
3. Presence of thrombus or suspected thrombus in the target vessel.
4. Aneurysm within 10 mm of the target lesion in the target vessel.
5. Presence of other lesions with stenosis >50% within the target vessel.
6. CTO lesion with excessive tortuosity (>45°) or length >20 mm.
7. Stent implanted within 5 mm proximal or distal to the target lesion.
8. Target lesion accessible only via saphenous vein graft (SVG) or arterial graft.
9. Failure of guidewire to successfully cross the target lesion.
10. Planned use of Antegrade Dissection Re-entry (ADR), Retrograde Wiring (RW), or Retrograde Dissection Re-entry (RDR) techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Device Success | immediately after IVL intervention
Freedom from Major Adverse Cardiovascular Events (MACE) within 30 days post-procedure | 30-day after the procedure

SECONDARY OUTCOMES:
Rate of Technical Success | immediately after the procedure
Rate of Angiographic Success | Peri-procedural
Rate of Procedural Success | at discharge/up to 7 days after the procedure
Incidence of serious angiographic complications | immediately after the procedure
Incidence of MACE | during procedure, at discharge (up to 7 days after the procedure) ,180 days after the procedure
Incidence of Target Lesion Failure | during procedure, at discharge (up to 7 days after the procedure), 30 days after the procedure, 180 days after the procedure
Incidence of Patient-Oriented Cardiovascular Endpoint | during procedure, at discharge (up to 7 days after the procedure), 30 days after the procedure, 180 days after the procedure
Incidence of Device Deficiencies | immediately after the prcedure
Excellent rate of device performance evaluation | Immediately after the procedure
Incidence of Adverse Events and Serious Adverse Events | through study completion, 180 days after the procedure

OTHER OUTCOMES:
Quantitative Coronary Angiography (QCA) Subgroup | immediately after the procedure
Optical Coherence Tomography (OCT) Subgroup | immediately after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China